CLINICAL TRIAL: NCT01471327
Title: A Single Blind, Placebo Controlled, Parallel Group, Single Ascending Intravenous Dose Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SB-240563 (Mepolizumab) in Healthy Japanese Male Subjects.
Brief Title: Japanese Phase 1 Study of Mepolizumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 115705
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — mepolizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- SB-240563, 10mg (Experimental): IV, single dose at Day 1
  Interventions: Biological: SB-240563
- Placebo (Experimental): Saline IV, single dose at Day 1
  Interventions: Other: Placebo
- SB-240563, 75mg (Experimental): IV, single dose at Day 1
  Interventions: Biological: SB-240563
- SB-240563, 250mg (Experimental): IV, single dose at Day 1
  Interventions: Biological: SB-240563
- SB-240563, 750mg (Experimental): IV, single dose at Day 1
  Interventions: Biological: SB-240563

INTERVENTIONS:
Biological: SB-240563 — 10mg, 75mg, 250mg and 750mg IV, single dose on Day 1
  Arms: SB-240563, 10mg; SB-240563, 250mg; SB-240563, 750mg; SB-240563, 75mg
Other: Placebo — Saline IV, single dose at Day 1
  Arms: Placebo

SUMMARY:
SB-240563 is a fully humanized monoclonal antibody which is specific for human interleukin-5 (IL-5) and has been under development for severe refractory asthma. This study is the first study in Japanese subjects. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single dose SB-240563 administered intravenously to Japanese healthy male subjects.

DETAILED DESCRIPTION:
Asthma is a disease characterised by chronic airway inflammation, bronchial hyper-reactivity and variable airflow obstruction. Eosinophils are usually prominent in the airway inflammation seen in asthma and are considered a central cause in the pathogenesis of asthma. The expression of interleukin (IL)-5 is elevated in bronchoalveolar lavage (BAL) fluid and bronchial biopsies in patients with asthma. Moreover, the level of IL-5 in BAL fluid and the bronchial mucosa correlates with disease severity. The cytokine IL-5 promotes eosinophil differentiation, recruitment and survival. Thus a therapeutic strategy which blocks IL-5, thereby suppressing eosinophilic inflammation, may have therapeutic benefit in asthma.

SB-240563 (mepolizumab) is a humanized monoclonal antibody that blocks human interleukin 5 (hIL-5) from binding to its receptor. Initial clinical studies investigated the safety and efficacy of SB-240563 for the treatment of asthma and atopic dermatitis (AD). SB-240563 consistently and significantly reduced peripheral and tissue eosinophils in patients with these atopic conditions, including asthma, and in healthy volunteers.

SB-240563 is currently under development for severe refractory asthma and a Phase IIB dose-ranging study using the IV route of administration is currently ongoing. This study will be a single-blind, placebo-controlled, parallel group, dose ascending, single dose study in Japanese healthy male subjects.

Since this is the first study conducted in Japanese subjects, doses of SB-240563 will be administered in an ascending order. In studies conducted in non-Japanese subjects, SB-240563 has been well-tolerated following single and repeated intravenous dose up to 750 mg (SB-240563/006, SB-240563/036 and MEE103226). Intravenous repeated doses of 75 mg, 250 mg and 750 mg are being administered to non-Japanese asthma patients in an on-going Phase II study. In consideration of the above facts, single intravenous administration of 4 doses (10 mg, 75 mg, 250 mg and 750 mg) of SB-240563 will be administered in this study. A single intravenous dose of 10 mg will be administered in order to explore the effect of a lower dose of SB-240563 than previously studied on blood eosinophil counts. This low dose is expected to help further characterize the concentration-response relationship based on blood eosinophils.

This study is designed as a randomized, parallel group, placebo-controlled, single-blind study to evaluate the pharmacokinetics, pharmacodynamics, safety and tolerability of SB-240563 in Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Japanese defined as being born in Japan, having four ethnic Japanese grandparents, holding a Japanese passport or identity papers and being able to speak Japanese. Japanese subjects should also have lived outside Japan for less than 10 years.
* Male between 20 and 55 years of age inclusive, at the time of signing the informed consent.
* Body weight equal or more than 45.0 kg and BMI within the range between 18.5 and 29.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* At screening, QTCF<450 msec; or QTcF < 480 msec in subjects with Bundle Branch Block.
* AST, ALT, alkaline phosphatase and bilirubin equal or less than 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:

an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units. One unit is equivalent to a 285 mL glass or full strength beer or 425 mL schooner or light beer or 1 (30 mL) measure of spirits or 1 glass (100 mL) of wine (NHMRC Guidelines [NHMRC, 2001])

* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Subjects with a smoking history of >10 cigarettes per day in the last 3 months.
* The subject's systolic blood pressure is outside the range of 90-140 mmHg, or diastolic blood pressure is outside the range of 45-90 mmHg or systolic blood pressure drop from supine to standing of >30 mmHg, or heart rate is outside the range of 40-100 bpm for subjects at Screening and pre-dose on Day 1.
* Exposure to live vaccine within the four weeks prior to screening or with intention to receive live vaccine during the study

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-08-09 (Actual); Primary Completion 2012-04-27 (Actual); Study Completion 2012-04-27 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics | From Day 1 to Follow-Up(Days 85 for Cohort 1 and 2, Days 121 for Cohort 3, Days 151 for Cohort 4)
  Cmax, AUC
Safety | From Day 1 to Follow-Up (Days 85 for Cohort 1 and 2, Days 121 for Cohort 3, Days 151 for Cohort 4)
  vital signs, ECGs, clinical laboratory tests and adverse events

SECONDARY OUTCOMES:
blood eosinophil counts | From Day 1 to Follow-Up (Days 85 for Cohort 1 and 2, Days 121 for Cohort 3, Days 151 for Cohort 4)
  change from baseline of blood eosinophils absolute counts
free and total IL5 levels | From Day 1 to Follow-Up (Days 85 for Cohort 1 and 2, Days 121 for Cohort 3, Days 151 for Cohort 4)
  Serum levels of free and total IL5
immunogenicity | From Day 1 to Follow-Up (Days 85 for Cohort 1 and 2, Days 121 for Cohort 3, Days 151 for Cohort 4)
  anti-SB-240563 antibody

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Clutterbuck EJ, Hirst EM, Sanderson CJ. Human interleukin-5 (IL-5) regulates the production of eosinophils in human bone marrow cultures: comparison and interaction with IL-1, IL-3, IL-6, and GMCSF. Blood. 1989 May 1;73(6):1504-12. PMID 2653458
- [Background] Haldar P, Brightling CE, Hargadon B, Gupta S, Monteiro W, Sousa A, Marshall RP, Bradding P, Green RH, Wardlaw AJ, Pavord ID. Mepolizumab and exacerbations of refractory eosinophilic asthma. N Engl J Med. 2009 Mar 5;360(10):973-84. doi: 10.1056/NEJMoa0808991. PMID 19264686
- [Background] Hamid Q, Azzawi M, Ying S, Moqbel R, Wardlaw AJ, Corrigan CJ, Bradley B, Durham SR, Collins JV, Jeffery PK, et al. Expression of mRNA for interleukin-5 in mucosal bronchial biopsies from asthma. J Clin Invest. 1991 May;87(5):1541-6. doi: 10.1172/JCI115166. PMID 2022726
- [Background] Humbert M, Corrigan CJ, Kimmitt P, Till SJ, Kay AB, Durham SR. Relationship between IL-4 and IL-5 mRNA expression and disease severity in atopic asthma. Am J Respir Crit Care Med. 1997 Sep;156(3 Pt 1):704-8. doi: 10.1164/ajrccm.156.3.9610033. PMID 9309982
- [Background] Robinson DS, Ying S, Bentley AM, Meng Q, North J, Durham SR, Kay AB, Hamid Q. Relationships among numbers of bronchoalveolar lavage cells expressing messenger ribonucleic acid for cytokines, asthma symptoms, and airway methacholine responsiveness in atopic asthma. J Allergy Clin Immunol. 1993 Sep;92(3):397-403. doi: 10.1016/0091-6749(93)90118-y. PMID 8360390
- [Background] Smith DA, Minthorn EA, Beerahee M. Pharmacokinetics and pharmacodynamics of mepolizumab, an anti-interleukin-5 monoclonal antibody. Clin Pharmacokinet. 2011 Apr;50(4):215-27. doi: 10.2165/11584340-000000000-00000. PMID 21348536
- [Background] Wang JM, Rambaldi A, Biondi A, Chen ZG, Sanderson CJ, Mantovani A. Recombinant human interleukin 5 is a selective eosinophil chemoattractant. Eur J Immunol. 1989 Apr;19(4):701-5. doi: 10.1002/eji.1830190420. PMID 2659368
- [Background] Wardlaw AJ, Brightling C, Green R, Woltmann G, Pavord I. Eosinophils in asthma and other allergic diseases. Br Med Bull. 2000;56(4):985-1003. doi: 10.1258/0007142001903490. PMID 11359633
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 115705 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115705?search=study&study_ids=115705#rs
- Available data/document: Annotated Case Report Form: 115705 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115705 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115705 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115705 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115705 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115705 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115705 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register